CLINICAL TRIAL: NCT02182973
Title: Donor Human Milk for Infants With Neonatal Abstinence Syndrome
Brief Title: Donor Human Milk in Neonatal Abstinence Syndrome
Acronym: DHM&NAS
Status: Completed | Type: Observational
Sponsor: Neolac Inc dba Medolac Laboratories (Industry)
Collaborators: University of Louisville (Other)
Responsible Party: Sponsor
Other Study IDs: NAS 052014
Record Dates: First submitted 2014-05-29; First posted 2014-07-08 (Estimated); Results first posted 2019-04-12 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Neonatal Abstinence Syndrome
Keywords: neonatal abstinence syndrome, infant opiate withdrawal
MeSH Terms: conditions — Neonatal Abstinence Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DHM: Infants identified with neonatal abstinence syndrome requiring pharmacologic management and who will not be fed own mother's milk
  Interventions: Dietary Supplement: donor human milk

INTERVENTIONS:
Dietary Supplement: donor human milk — Infants with NAS requiring pharmacologic management will be fed donor human milk instead of formula for 2 weeks.
  GI-subscores from the Finnegan NAS Scoring system will be computed.
  Other Names: Co-op donor milk (Medolac Laboratories)

SUMMARY:
This study is designed to develop pilot data on the acceptability and benefit of donor human milk for infants undergoing pharmacologic treatment for NAS. Specifically, gastrointestinal (GI) sub-scores, as well as total scores, will be compared between infants historically fed formula and those enrolled in a 2-week donor human milk study period.

Purpose of study: to test the following null hypothesis:

Infants with a diagnosis of neonatal abstinence syndrome (NAS) due to in-utero exposure to opiates, fed donor human milk, will have similar GI/feeding sub-scores of the Finnegan scoring tool when compared to (historic) infants fed formula.

A rejection of the null hypothesis will be used to design a randomized trial of donor human milk in infants with NAS.

DETAILED DESCRIPTION:
Background

Neonatal Abstinence Syndrome (NAS) is a drug withdrawal syndrome that occurs primarily after antenatal exposure to opiates. Symptoms may be present at birth, but often peak at 48-72 after delivery. The onset of symptoms is affected by the half-life of the opiate used during pregnancy in combination with maternal and infant metabolism. The incidence of NAS has increased substantially since 2000 both nationally and in the Commonwealth of Kentucky, leading to a significant increase in healthcare resource utilization and (Figure 1).

The 2012 National Survey on Drug Use and Health found that illicit drug abuse affected ~130,000 pregnancies in the United States from 2011-2012 and that approximately 20% of those pregnancies (26,000) involved opiates. (SAMSA Center for Behavioral Health Statistics and Quality, National Survey on Drug Use and Health, 2009-2012). Patrick et al. utilized the Kids' Inpatient Database (KID) from the Agency for Health Care Research and Quality to evaluate the incidence of maternal opiate use during pregnancy (1). He and his team noted a substantial increase in the number of mothers using opiates - 1.19 per 1000 hospital births in 2000 to 5.63 per 1000 hospital births in 2009. As a result, there was an increased diagnosis of NAS from 1.20 per 1000 hospital births in 2000 to 3.39 per 1000 hospital births in 2009. This is a 2.8-fold increase which means that every hour of every day, 1 neonate in the United States undergoes drug withdrawal.

The Kentucky Injury Prevention and Research Center reported that 824 infants in the state of Kentucky were hospitalized for neonatal withdrawal after exposure to opiates in 2012. This represents an 18% increase from 2011 and a 4.5 fold increase from 2005. (Kentucky Injury Prevention and Research Center. Data for 2010-2012). NAS is an issue of epidemic proportions both for Kentucky and the nation. It results in prolonged hospitalizations and increased healthcare costs. In 2009, the total charges for NAS treatment were noted to be approximately $720 million nationally, up from approximately $190 million in 2000 (1). Kentucky data from 2012 report a $40 million dollar cost for neonatal drug withdrawal treatment, which has increased from $200,000 in 2000. (Kentucky Injury Prevention and Research Center. Data for 2010-2012). The majority of these costs (75-80%) are paid by the state Medicaid program (Figure 2).

Precipitous removal of exogenous opiates at the time of delivery results in unopposed stimulation by cyclic adenosine monophosphate (cAMP) and which increases norepinephrine levels and results in clinical symptoms of drug withdrawal in the neonate (2). Symptoms include central nervous system (CNS) signs (seizures, irritability, tremors), autonomic disturbances (sweating, yawning, nasal stuffiness, low grade fever, mottling) and gastrointestinal (GI) dysfunction (diarrhea, vomiting, poor feeding, and regurgitation). The cohort of withdrawal symptoms is dictated by the location of µ opioid receptors, which are concentrated in the brain but are also found in sensory nerves, mast cells and in the GI tract(3).

Treatment of withdrawal symptoms includes symptomatic care for mild symptoms and pharmacological intervention in addition to symptomatic care for moderate to severe symptoms. The American Academic of Pediatrics (AAP) and experts in the field recommend opioid replacement therapy as the first line pharmacologic intervention in opioid-induced withdrawal. The most commonly used medication is oral morphine. Phenobarbital and clonidine have been used as adjuvant therapies with some success in infants with more severe symptoms. Initiation, escalation and weaning of pharmacologic therapy are based on observer rated scales, the most common of which is the Finnegan Scale(4). Although observer-rated scales are an essential component in the assessment and treatment of neonatal drug withdrawal, they lack rigorous psychometric testing to establish reliability and validity, are subjective and have been difficult to standardize across nurseries (5).

Infants undergoing opiate withdrawal, as noted above, have feeding difficulty, including spitting, regurgitation and diarrhea. The Finnegan scoring tool includes a series of feeding assessments within the total scoring algorithm (Table 1). Human milk has been shown to be the best tolerated nutritional support for most infants and is cited by the AAP as the preferred method for feeding all infants (6). However, the AAP considers the use of marijuana, cocaine, methamphetamines and unsupervised opiate use during pregnancy to be a contraindication to breastfeeding (7). For most street drugs, the risks to the infant of ongoing active use by the mother outweigh the benefits of breastfeeding because the doses of the drug(s) being used and contaminants within the drug are unknown (8-11). The AAP does recognize that if a mother is in a supervised methadone treatment center and is free from using other drugs of abuse then breastfeeding is an essential component of the infant's care. However, most infants with NAS are fed formula for a variety of reasons, including concerns about continued maternal use.

Human milk is a complete nutritional food for the first 6 months of life in the term infant. Aside from its nutritional composition (specific for the support of the human infant), it contains hormones, immunoglobulins and growth factors that stimulate gastrointestinal growth and motility which, in turn, promote the maturation and protection of the GI tract. Mediators such as neurotensin and motilin promote GI motility while free amino acids feed intestinal growth (12,13). Human milk feeding has been shown to increase gastric emptying (14,15) and lactase activity (16) in the gut which improves feeding tolerance. A human milk diet is also associated with post-natal intestinal colonization by beneficial bacteria (Lactobacillus and Bifidobacteria). In summary, when compared to formula feeding, human milk appears to be a more suitable diet for the neonate at risk for GI dysfunction.

Two retrospective studies of the effect of breastfeeding on clinical symptoms of NAS have been reported. McQueen et al reviewed 28 mother-infant pairs with maternal methadone exposure and infant symptoms of NAS (17). Maternal and infant demographics were recorded along with feeding type, Finnegan scores and infant medication utilization during withdrawal. Feeding cohorts were created by quantifying the duration of breastfeeding during hospitalization. Formula fed infants received >75% of all feedings as formula (n=9), breastfed infants received >75% of feedings at the breast (n=8). The rest were considered combination feeders (n=11). Combination feeders were slightly less mature (35.6 weeks) and of lower birth weight (2608 g) than breastfed (38.8 weeks and 3025 g) or formula fed (39.1 weeks and 3302 grams). Breastfed infants received fewer scores, had significantly lower overall Finnegan scores and fewer scores >8 when compared to formula and combination fed infants (p≤0.001).

Dryden et al. performed a retrospective cohort study of 437 infants born to women prescribed methadone in varying doses for their addiction (18). Median gestational age at birth was 38 weeks and birth weight was 2730 grams. Twenty-two percent of infants were breastfed for at least 72 hours. Multivariate logistic regression showed that the prescribed dose of methadone in these women independently influenced the likelihood of pharmacologic treatment for NAS (p<0.001). However, for infants that were breastfed for at least 72 hours, the odds of needing pharmacologic treatment for NAS was significantly reduced (OR 0.55, 95% confidence interval 0.34 - 0.88, p=0.013).

Maternal opiates are transmitted through the breast milk to the infant. The amount of methadone and buprenorphine transferred in the breast milk has been found to be small, but may be significant enough to lead to some improvement in scores.

While these studies have reported improvements (decreases) in NAS scoring or reduced duration of treatment with breastfeeding, there are no reports that have looked at donor human milk, which is tested to be free of illicit drugs, and its effect on the GI sub-scores of the Finnegan algorithm. Given the general benefits of human milk for the human infant and these limited reports of improved neonatal well-being in breastfed infants with NAS, this study is designed to develop pilot data on the acceptability and benefit of donor human milk for infants undergoing pharmacologic treatment for NAS. Specifically, GI sub-scores, as well as total scores, will be compared between infants historically fed formula and those enrolled in a 2-week donor human milk study period.

Purpose of study: to test the following null hypothesis:

Infants with a diagnosis of neonatal abstinence syndrome (NAS) due to in-utero exposure to opiates, fed donor human milk, will have similar GI/feeding sub-scores of the Finnegan scoring tool when compared to (historic) infants fed formula.

A rejection of the null hypothesis will be used to design a randomized trial of donor human milk in infants with NAS.

Methods:

Once the infant's withdrawal symptoms have been stabilized with oral morphine and the mother has agreed to participation (signed informed consent and research authorization), infants will be assigned to receive only donor human milk (Co-op donor milk, Medolac Laboratories, Lake Oswego, OR) for a period of 2 weeks. Vitamin supplementation or other nutritional adjustments will be at the discretion of the attending physician.

Infant Finnegan scores will be assessed according to the current NAS protocol. Oral morphine dosing (increases or weaning doses) will be consistent with the current NAS protocol.

See data collection sheet for detailed list of variables.

Statistical analysis:

Descriptive statistics will be provided. As this is a pilot study, no inferential statistics will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Term infants (>37 completed weeks) with a diagnosis of NAS, due to maternal use of opiates (only)
* Infants will have had moderate to severe NAS symptoms (Finnegan scores >8) that required pharmacologic therapy but have been stabilized (captured) on oral morphine (Finnegan scores less than 8 for 24 hours)
* Breastfeeding is contraindicated or the mother has chosen formula feeding for her baby

Exclusion Criteria:

* Preterm infants (<37 completed weeks at birth)
* Infants with intrauterine growth restriction (BW <10th percentile for gestational age)
* Mother is providing her own milk

Ages: 38 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants with a diagnosis of neonatal abstinence syndrome (NAS) due to in-utero exposure to opiates, fed donor human milk, will have similar GI/feeding sub-scores of the Finnegan scoring tool when compared to (historic) infants fed formula.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori Devlin, DO, MHA, Principal Investigator — University of Louisville Division of Neonatal Medicine; Paula G Radmacher, MSPH, Ph.D., Study Director — University of Louisville Division of Neonatal Medicine; Scott Duncan, MD, Principal Investigator — University of Louisville Division of Neonatal Medicine
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Patrick SW, Schumacher RE, Benneyworth BD, Krans EE, McAllister JM, Davis MM. Neonatal abstinence syndrome and associated health care expenditures: United States, 2000-2009. JAMA. 2012 May 9;307(18):1934-40. doi: 10.1001/jama.2012.3951. Epub 2012 Apr 30. PMID 22546608
- [Background] Nestler EJ. Molecular mechanisms of opiate and cocaine addiction. Curr Opin Neurobiol. 1997 Oct;7(5):713-9. doi: 10.1016/s0959-4388(97)80094-3. PMID 9384550
- [Background] Kreek MJ, Bart G, Lilly C, LaForge KS, Nielsen DA. Pharmacogenetics and human molecular genetics of opiate and cocaine addictions and their treatments. Pharmacol Rev. 2005 Mar;57(1):1-26. doi: 10.1124/pr.57.1.1. PMID 15734726
- [Background] Kron RE, Finnegan LP, Kaplan SL, Litt M, Phoenix MD. The assessment of behavioral change in infants undergoing narcotic withdrawal: comparative data from clinical and objective methods. Addict Dis. 1975;2(1-2):257-75. PMID 1163368
- [Background] Neonatal drug withdrawal. American Academy of Pediatrics Committee on Drugs. Pediatrics. 1998 Jun;101(6):1079-88. PMID 9614425
- [Background] Section on Breastfeeding. Breastfeeding and the use of human milk. Pediatrics. 2012 Mar;129(3):e827-41. doi: 10.1542/peds.2011-3552. Epub 2012 Feb 27. PMID 22371471
- [Background] Behnke M, Smith VC; Committee on Substance Abuse; Committee on Fetus and Newborn. Prenatal substance abuse: short- and long-term effects on the exposed fetus. Pediatrics. 2013 Mar;131(3):e1009-24. doi: 10.1542/peds.2012-3931. Epub 2013 Feb 25. PMID 23439891
- [Background] Chasnoff IJ, Lewis DE, Squires L. Cocaine intoxication in a breast-fed infant. Pediatrics. 1987 Dec;80(6):836-8. PMID 3684393
- [Background] COBRINIK RW, HOOD RT Jr, CHUSID E. The effect of maternal narcotic addiction on the newborn infant; review of literature and report of 22 cases. Pediatrics. 1959 Aug;24(2):288-304. No abstract available. PMID 13674828
- [Background] Perez-Reyes M, Wall ME. Presence of delta9-tetrahydrocannabinol in human milk. N Engl J Med. 1982 Sep 23;307(13):819-20. doi: 10.1056/NEJM198209233071311. No abstract available. PMID 6287261
- [Background] Steiner E, Villen T, Hallberg M, Rane A. Amphetamine secretion in breast milk. Eur J Clin Pharmacol. 1984;27(1):123-4. PMID 6489423
- [Background] Rodriguez-Palmero M, Koletzko B, Kunz C, Jensen R. Nutritional and biochemical properties of human milk: II. Lipids, micronutrients, and bioactive factors. Clin Perinatol. 1999 Jun;26(2):335-59. PMID 10394491
- [Background] Sheard NF, Walker WA. The role of breast milk in the development of the gastrointestinal tract. Nutr Rev. 1988 Jan;46(1):1-8. doi: 10.1111/j.1753-4887.1988.tb05343.x. No abstract available. PMID 3277089
- [Background] Billeaud C, Guillet J, Sandler B. Gastric emptying in infants with or without gastro-oesophageal reflux according to the type of milk. Eur J Clin Nutr. 1990 Aug;44(8):577-83. PMID 2209513
- [Background] Cavell B. Gastric emptying in infants fed human milk or infant formula. Acta Paediatr Scand. 1981 Sep;70(5):639-41. PMID 7324911
- [Result] Alexander C, Radmacher P, Devlin L. Donor human milk may decrease severe gastrointestinal distress in infants with neonatal abstinence syndrome. Pregnancy and neonatal medicine 2017; 1(1):11-15.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Historical controls are not considered to be enrolled in the study. Thus, they are not counted in the enrollment numbers.
Groups:
- Donor Human Milk: Infants identified with neonatal abstinence syndrome requiring pharmacologic management and who will not be fed own mother's milk
  donor human milk: Infants with NAS requiring pharmacologic management will be fed donor human milk instead of formula for 2 weeks.
  GI-subscores from the Finnegan NAS Scoring system will be computed.
- Historical Control: Infants from the previous year with NAS but fed formula.
Period: Overall Study
Arm/Group | Donor Human Milk | Historical Control
Started | 12 | 9
Completed | 9 | 9
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Population: 1. Infants with a diagnosis of neonatal abstinence syndrome (NAS) and
  2. The mother had elected formula for the infant's feeding.
Groups:
- Donor Human Milk: Term infants identified with neonatal abstinence syndrome requiring pharmacologic management and who will not be fed own mother's milk
  Donor human milk: Infants with NAS requiring pharmacologic management will be fed donor human milk instead of formula for 2 weeks.
  GI-subscores from the Finnegan NAS Scoring system will be computed.
- Historical Control: Term infants identified with NAS requiring pharmacologic management in the previous year receiving formula feedings.
- Total: Total of all reporting groups
Arm/Group | Donor Human Milk | Historical Control | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants] — Gestational age by neonatologist's estimate or obstetrical history Population: 3 subjects were withdrawn by a parent prior to completing the study.
  Participants
    <=18 years | 9 | 9 | 18
    Between 18 and 65 years | 0 | 0 | 0
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 38.8 (1.0) | 38.8 (1.4) | 38.8 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 7 | 5 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 0 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 9 | 9
Region of Enrollment [Count of Participants; unit: Participants] — Population: 3 infants were withdrawn from the study by the parent early in the study and were not in the final analyzed group.
  Participants
    United States | 9 | 9 | 18
Birth weight [Mean (Standard Deviation); unit: grams] | 3091 (350) | 2934 (495) | 3013 (423)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Infants Achieving a GI Subscore >2 Over the Study Period
Description: Minimum score:0; Maximum score 13. Higher scores mean more GI distress
Time Frame: 2 weeks
Measure: Number; unit: Percentage of participants
Groups:
- Historical Controls: Historical groups with NAS and receiving formula
Arm/Group | Donor Human Milk | Historical Controls
Number analyzed (Participants) | 9 | 9
Percentage of participants | 39 | 61
Statistical Analysis 1: Comparison: Donor Human Milk vs Historical Controls; Test type: Superiority; p = 0.001, t-test, 2 sided

2. Secondary Outcome: Weight Change at 2 Weeks
Description: Change in weight from study day 1 to study day 14 (grams/day) Weight day 14 - weight day 1 divided by 14
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: grams/day
Groups:
- Historical Control: Historical groups with NAS and receiving formula
Arm/Group | Donor Human Milk | Historical Control
Number analyzed (Participants) | 9 | 9
grams/day | 19.1 (13.1) | 20.5 (3.0)
Statistical Analysis 1: Comparison: Donor Human Milk vs Historical Control; Test type: Superiority; p = 0.875, t-test, 2 sided

3. Secondary Outcome: Head Circumference Change at 2 Weeks
Description: Change in head circumference from day 1 to day 14 (cm/wk)
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: cm/wk
Arm/Group | Donor Human Milk | Historical Control
Number analyzed (Participants) | 9 | 9
cm/wk | 0.4 (0.1) | 0.6 (0.2)
Statistical Analysis 1: Comparison: Donor Human Milk vs Historical Control; Test type: Superiority; p = 0.025, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Study period (2 weeks)
Description: For the historical control group, adverse events were monitored per standard of care.
Arm/Group | Donor Human Milk | Historical Control
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/9
Other Adverse Events (participants affected / at risk) | 0/12 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-05-09): https://cdn.clinicaltrials.gov/large-docs/73/NCT02182973/Prot_SAP_000.pdf